CLINICAL TRIAL: NCT01859520
Title: The Effect of Swim up and Gradient Methods Used in Assisted Reproduction Techniques on DNA Fragmentation of Spermatozoa
Brief Title: Swim up and Gradient Methods Used in Assisted Reproduction Techniques on DNA Fragmentation of Spermatozoa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Prof Ahmet ERDEM, MD, Professor of Obstetrics and Gynecology, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gazi University 01/2011-110
Record Dates: First submitted 2013-03-25; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Male Infertility; Unexplained Infertility
Keywords: Spermatozoa; DNA fragmentation; Swim-up; Density gradient
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Swim up, density gradient (Experimental): swim-up and density gradient sperm preparation techniques in male factor infertility and unexplained infertility groups
  Interventions: Procedure: swim-up, density gradient sperm preparation techniques

INTERVENTIONS:
Procedure: swim-up, density gradient sperm preparation techniques — Sperms are prepared by sperm washing techniques before used in assisted reproductive technologies. Most commonly used sperm preparation methods are the swim up and the density gradient. Recent studies shows that the DNA integrity status of the spermatozoa is related to the success in assisted reproduction techniques. Sperm preparation methods may theoretically cause damage sperm DNA. Therefore it is important to select the optimum method of sperm preparation causing least sperm DNA damage. Aim of our study is to investigate and compare the effect two different sperm preparation techniques on DNA fragmentation.

SUMMARY:
Sperms are prepared by sperm washing techniques before used in assisted reproductive technologies. Most commonly used sperm preparation methods are the swim up and the density gradient. Recent studies shows that the DNA integrity status of the spermatozoa is related to the success in assisted reproduction techniques. Sperm preparation methods may theoretically cause damage to sperm DNA. Therefore it is important to select the optimum method of sperm preparation causing least sperm DNA damage. Aim of our study is to investigate and compare the effect two different sperm preparation techniques on DNA fragmentation.

ELIGIBILITY:
Inclusion Criteria:

Male factor subfertile group:

Couples of having at least two abnormal sperm analysis according to WHO criteria.

Unexplained subfertile group:

Couples with normal sperm parameters, plus females with normal ovulatory status and patent fallopian tubes by hysterosalpingography or laparoscopy.

No previous IVF or IUI attempts before the study

Exclusion Criteria:

Severe oligospermia (Sperm count < 5 Millions/ per ml) Systemic diseases or therapies influencing DNA integrity for male partner

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The change in the rate of DNA fragmentation of spermatozoa after sperm preparation with either swim-up or density gradient techniques. | DNA fragmentation assay is performed just before and immediately after the sperm preparation is completed. The time frame is within an hour.
  The change in the rate of DNA fragmented spermatozoa will be assessed before and immediately after the sperm preparation is completed, because DNA fragmentation of spermatozoa may be increased in time.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet erdem, Professsor, MD, Study Director — University of Gazi School of Medicine Department of Obstetrics and Gynecology; Yuksel Oguz, Resident, MD, Principal Investigator — University of Gazi School Of Medicine Department of Obstetrics and Gynecology